CLINICAL TRIAL: NCT04630223
Title: Comparison of Umbilical Cord Blood Levels of Endocan in Pregnant Females With and Without Intrauterine Growth Retardation
Brief Title: Levels of Endocan in Umbilical Cord Blood Samples of Pregnant Females With Intrauterine Growth Retardation
Status: Completed | Type: Observational
Sponsor: Van Bölge Eğitim ve Araştırma Hastanesi (Other Government)
Responsible Party: Principal Investigator, cagdas özgökce, MD, specialist on obstetrics and gynecology, Van Bölge Eğitim ve Araştırma Hastanesi
Other Study IDs: EndocanIUGR
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Intrauterine Retardation
Keywords: intrauterine growth retardation; umbilical cord blood; proteoglycans; pregnancy outcomes
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intrauterine growth retardation: Blood samples are going to be taken from the umbilical cord of the fetuses. Levels of endocan (endothelial cell specific molecule 1) in the samples of umbilical cord blood are going to be measured using human endocan ELISA kits.
  Interventions: Diagnostic Test: endocan in umbilical cord blood
- healthy fetuses: Blood samples are going to be taken from the umbilical cord of healthy fetuses without intrauterine growth retardation. Levels of endocan (endothelial cell specific molecule 1) in the samples of umbilical cord blood are going to be measured using human endocan ELISA kits.
  Interventions: Diagnostic Test: endocan in umbilical cord blood

INTERVENTIONS:
Diagnostic Test: endocan in umbilical cord blood — After taking blood samples from the umbilical cord, centrifugation is applied to all samples for 15 minutes at 1000 rpm. The serum samples with specific identification numbers are going to be stored at -80 °C. After completing the study group, all serum samples will be analyzed using human endocan ELISA kit for the measurement of endocan levels.

SUMMARY:
As a proteoglycan secreted from endothelial cells, expression, and secretion of endocan increases in the endothelium of several tissues secondary to inflammation. It can be regarded as an indicator of endothelial damage. Besides, it is both a target and a modulator of the vascular endothelial growth factor (VEGF) signaling pathway. Considering its action mechanisms, it can provide information about angiogenesis, inflammation, and vascular permeability.

It is known that intrauterine growth retardation mainly occurs as a result of endothelial dysfunction and abnormal angiogenesis in the placenta. In previous studies, maternal serum endocan levels have also been shown to be increased in cases of preeclampsia, which is mainly characterized by placental dysfunction.So, we hypothesize that there may be an association between endocan levels and intrauterine growth retardation.

DETAILED DESCRIPTION:
Endocan is a proteoglycan that is closely associated with inflammation. Its levels increase in association with the severity of endothelial damage. Endothelial dysfunction and abnormal angiogenesis in the placental tissues are the main pathophysiological mechanisms leading to intrauterine growth retardation.

It has been known that there was a significant association between maternal serum levels of endocan and preeclampsia. In cases with preeclampsia, increased serum levels of endocan in maternal blood samples has been reported.

Intrauterine growth retardation is a situation in which endothelial dysfunction and abnormal angiogenesis are the leading disturbances. In fetuses with intrauterine growth retardation, a hypoxic environment secondary to uteroplacental insufficiency. In previous studies, increased levels of endocan in maternal blood samples have been shown. Although maternal blood can be a good reflector of situations both in fetuses and their mothers, measurement of endocan in umbilical cord blood samples may better represent the pathology in fetuses.

ELIGIBILITY:
Inclusion Criteria:

For "intrauterine growth retardation" group:

* consent to participate study
* detection of intrauterine growth retardation during follow up of pregnancy

For "healthy fetuses" group:

* consent to participate study
* absence of intrauterine growth retardation during follow up of pregnancy

Exclusion Criteria:

* multiple pregnancy
* presence of major developmental anomalies of fetuses
* detection of chromosomal anomalies
* malnourished mothers
* vegetarian diet of mothers
* use of cigarette and alcohol during pregnancy
* previous history of stillbirths

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female pregnants
Study Population: Pregnant females attending outpatient clinics of obstetrics in a tertiary hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
endocan in umbilical cord blood | just after delivery of fetus at clamping of umbilical cord
  levels of endothelial cell specific molecule 1 (ng/ml) in umbilical cord blood

CONTACTS AND LOCATIONS:
Locations (1):
- Van Region Education and Training Hospital, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Medical data of the participants are going o be shared if it is requested.

REFERENCES:
- [Result] Kucukbas GN, Kara O, Yuce D, Uygur D. Maternal plasma endocan levels in intrauterine growth restriction. J Matern Fetal Neonatal Med. 2022 Apr;35(7):1295-1300. doi: 10.1080/14767058.2020.1749591. Epub 2020 Apr 14. PMID 32290736
- [Result] Lan X, Liu Z. Circulating endocan and preeclampsia: a meta-analysis. Biosci Rep. 2020 Jan 31;40(1):BSR20193219. doi: 10.1042/BSR20193219. PMID 31854443
- [Result] Szpera-Gozdziewicz A, Kosicka K, Gozdziewicz T, Krzyscin M, Wirstlein P, Siemiatkowska A, Glowka F, Wender-Ozegowska E, Breborowicz GH. Maternal Serum Endocan Concentration in Pregnancies Complicated by Intrauterine Growth Restriction. Reprod Sci. 2019 Mar;26(3):370-376. doi: 10.1177/1933719118773480. Epub 2018 May 9. PMID 29742984